CLINICAL TRIAL: NCT02332798
Title: A Randomized, Double-blind, Placebo Controlled, Sponsor Open, Parallel Group Phase 1b Study To Examine The Safety, Tolerability And Pharmacokinetics Of Multiple Ascending Doses Of Pf-04958242 In Subjects With Stable Schizophrenia
Brief Title: Multiple Ascending Doses of PF-04958242 in Subjects With Stable Schizophrenia
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1701017; MAD (Other: Alias Study Number)
Record Dates: First submitted 2014-12-05; First posted 2015-01-07 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Schizophrenia
Keywords: Multiple ascending doses; safety; tolerability; pharmacokinetics; cognitive impairment associated with schizophrenia (CIAS)
MeSH Terms: conditions — Schizophrenia | interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-04958242 0.25 mg (Experimental): All participants who received PF-04958242 0.25 milligram (mg) twice daily (BID) for 14 consecutive days with the last dose occurring in the morning on Day 14.
  Interventions: Drug: PF-04958242
- PF-04958242 0.475 mg (Experimental): All participants who received PF-04958242 0.475 mg BID for 14 consecutive days with the last dose occurring in the morning on Day 14.
  Interventions: Drug: PF-04958242
- Matching Placebo (Placebo Comparator): All participants who received placebo BID for 14 consecutive days with the last dose occurring in the morning on Day 14.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04958242 — Administered as specified in the treatment arm
  Arms: PF-04958242 0.25 mg; PF-04958242 0.475 mg
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Matching Placebo

SUMMARY:
This study aims to assess the safety, tolerability and pharmacokinetics of PF-04958242 in multiple ascending doses in subjects with stable schizophrenia.

DETAILED DESCRIPTION:
This study aims to assess the safety, tolerability and pharmacokinetics of PF-04958242 compared to placebo over 14 days twice a day dosing in multiple ascending doses in subjects with stable schizophrenia.

This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Psychiatrically stable (≥3 months) male and female subjects with schizophrenia of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >55 kg (121 lbs).
* DSM-IV Diagnosis of Schizophrenia; on stable medication treatment regimen ≥2 months.

Key Exclusion Criteria:

* Suicide attempt within 3 months prior to screening.
* History of or risk of seizures; head injury with long term abnormal resulting condition, abnormal EEG, clinically significant additional diseases or conditions, current medication with a significant risk of seizures, currently receiving antipsychotic medications.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Collaborative Neuroscience Network, LLC., Long Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: All participants who received placebo BID for 14 consecutive days with the last dose occurring in the morning on Day 14.
Period: Overall Study
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Started | 13 | 14 | 12
Completed | 12 | 12 | 11
Not Completed | 1 | 2 | 1
Not completed — Unwilling to Participate in Study | 0 | 1 | 1
Not completed — Positive Urine Drug Test | 0 | 1 | 0
Not completed — Abnormal Laboratory Findings | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-04958242 0.25 mg: All participants who received PF-04958242 0.25 mg BID for 14 consecutive days with the last dose occurring in the morning on Day 14.
- Total: Total of all reporting groups
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo | Total
Number analyzed (Participants) | 13 | 14 | 12 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (5.9) | 41.6 (7.5) | 45.8 (10.5) | 44.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 5
  Male | 13 | 11 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) (Single Dose)
Time Frame: Day 1 (0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, and 12 hours post-dose)
Population: The pharmacokinetic (PK) concentration population is defined as all enrolled subjects treated who received at least one dose of PF-04958242 and have at least 1 measureable concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 13 | 14
nanograms per milliliter (ng/mL) | 1.920 (23) | 3.830 (21)

2. Primary Outcome: Cmax (Steady State)
Description: Cmax steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: Day 1 (0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12 hours post-dose), Day 2, Day 7 (0, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12 hours post-dose), Day 8, Day 10, Day 14 (0, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12 hours post-dose), Day 15, Day 17, Day 21
Population: The PK concentration population is defined as all enrolled subjects treated who received at least one dose of PF-04958242 and have at least 1 measureable concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 3.174 (18) | 7.139 (37)

3. Primary Outcome: Time for Cmax (Tmax) (Single Dose)
Time Frame: Day 1 (0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, and 12 hours post-dose)
Population: The PK analysis population included all participants enrolled and treated who had at least 1 of the PK parameters interest measured.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 13 | 14
hours | 1.65 [1.00 to 2.00] | 1.33 [0.167 to 3.00]

4. Primary Outcome: Tmax (Steady State)
Description: Tmax steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
hours | 1.65 [1.00 to 2.00] | 1.33 [0.50 to 4.00]

5. Primary Outcome: Area Under the Concentration-Time Profile From Time 0 to Time Tau (τ), the Dosing Interval, Where τ = 12 Hours (AUCτ) (Single Dose)
Time Frame: Day 1 (0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, and 12 hours post-dose)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 13 | 14
nanograms*hours per milliliter (ng*h/mL) | 9.570 (19) | 17.72 (18)

6. Primary Outcome: AUCτ (Steady State)
Description: AUCτ steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
ng*h/mL | 24.57 (19) | 50.09 (34)

7. Primary Outcome: Apparent Oral Clearance (CL/F) (Steady State)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute (mL/min)
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
milliliter per minute (mL/min) | 169.5 (18) | 157.9 (34)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F) (Steady State)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. Vz/F steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
Liter (L) | 545.7 (31) | 530.2 (26)

9. Primary Outcome: Terminal Half-Life (t1/2) (Steady State)
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half. t1/2 steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
hours | 39.64 (14.878) | 42.18 (14.421)

10. Primary Outcome: Observed Accumulation Ratio (Rac) (Steady State)
Description: Accumulation ratio was calculated as, Rac obtained from Area Under the Concentration Time Curve (AUC) from time 0-t (Day X) divided by AUC from time 0-t (Day 1). Rac steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 (ie. X = 14) were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
Ratio | 2.524 (20) | 2.815 (31)

11. Primary Outcome: Observed Accumulation Ratio for Cmax (Rac, Cmax) (Steady State)
Description: Accumulation ratio based on Cmax was calculated as: Rac,Cmax = Cmax at steady state (ss) divided by Cmax at first dose. Rac, Cmax steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
Ratio | 1.645 (23) | 1.797 (51)

12. Primary Outcome: Peak-to-Trough Ratio at Steady State (PTR)
Description: PTR was calculated as Cmax divided by Cmin (that is defined as lowest concentration observed during the dosing interval). PTR steady state for PF-04958242 0.25 mg group and PF-04958242 0.475 mg group at Day 14 were presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg
Number analyzed (Participants) | 12 | 12
Ratio | 2.323 (19) | 2.531 (28)

13. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Measurements
Description: The following laboratory parameters were reported: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], mean corpuscular hemoglobin concentration [MCHC], platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, phosphorus, cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), bicarbonate, uric acid, albumin, and total protein); urinalysis (color, appearance, specific gravity, pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, and microscopy); others (follicle stimulating hormone [FSH], and urine drug screening).
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 12
participants | 4 | 4 | 7

14. Primary Outcome: Number of Participants With Vital Signs Data Meeting Criteria of Potential Clinical Concern
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate less than (<) 40 or greater than (>) 120 beats per minute (bpm), standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from baseline in same posture or SBP <90 mm Hg, diastolic blood pressure (DBP) >=20 mm Hg change from baseline in same posture or DBP <50 mm Hg. IFB = increase from baseline; DFB = decrease from baseline.
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 12
participants
  Supine SBP <90 mmHg | 0 | 2 | 0
  Standing SBP <90 mmHg | 0 | 1 | 0
  Supine SBP >=30 mmHg IFB | 0 | 0 | 1
  Standing SBP >=30 mmHg IFB | 2 | 1 | 1
  Supine DBP >=20 mmHg IFB | 0 | 2 | 1
  Standing DBP >=20 mmHg IFB | 2 | 2 | 0
  Supine SBP >=30 mmHg DFB | 2 | 1 | 0
  Standing SBP >=30 mmHg DFB | 2 | 1 | 1
  Supine DBP >=20 mmHg DFB | 2 | 0 | 3
  Standing DBP >=20 mmHg DFB | 5 | 2 | 4

15. Primary Outcome: Number of Participants With Electrocardiogram Data Meeting Criteria of Potential Clinical Concern
Description: Electrocardiogram (ECG) parameters included beginning of the P wave until the beginning of the QRS complex (PR) interval, time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS) interval, and QTc using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval >=300 milliseconds (msec) or >=25% increase when baseline is >200 msec and >=50% increase when baseline is less than or equal to (=<)200 msec; QRS interval >=140 msec or >=50% increase from baseline (IFB); and and QTcF >=450 to <480, 480 to <500 and >=500 msec. The number of participants with potentially clinically significant ECG findings at any visit were reported.
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 12
participants | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Abnormalities in Neurological Examination
Description: The extended neurological examination, performed by a board certified neurologist, included observation for cerebellar (intention) tremor and for non-cerebellar tremors (eg, resting or positional), finger, nose, heel, shin, Romberg, tandem walking, positional and gaze evoked nystagmus, reflexes, muscle strength, cranial nerves, sensory function of upper and lower extremities. The brief neurological examination included an assessment of motor and sensory function, cranial nerves, reflexes, non-cerebellar tremor (eg, resting or positional) and cerebellar function. The assessment of cerebellar function were complemented by the Scale for Assessment and Rating of Ataxia (SARA).
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 12
participants | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Abnormalities in Physical Examination
Description: A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The brief physical examination focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms.
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 12
participants | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after last study drug administration
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 12
participants
  AEs | 10 | 9 | 4
  SAEs | 0 | 0 | 0

19. Primary Outcome: Number of Participants With Positive Response to Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced the following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 12
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration.
Arm/Group | PF-04958242 0.25 mg | PF-04958242 0.475 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 10/13 | 9/14 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04958242 0.25 mg (N=13) | PF-04958242 0.475 mg (N=14) | Placebo (N=12)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0
Nodule (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 4 | 4 | 2
Somnolence (Nervous system disorders) | 3 | 2 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.